CLINICAL TRIAL: NCT06572618
Title: A Phase 2 Study of BTK Inhibitor Nemtabrutinib in Combination With Rituximab in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: Nemtabrutinib With Rituximab for the Treatment of Patients With Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23421; NCI-2024-06740 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23421 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Specimen Handling; Biopsy; ARQ531; Magnetic Resonance Spectroscopy; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nemtabrutinib and rituximab) (Experimental): INDUCTION: Patients receive nemtabrutinib PO QD on days 1-28 of each cycle and rituximab IV on days 1, 8, 15 and 22 of cycle 1 and on day 1 of subsequent cycles. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive nemtabrutinib PO QD on days 1-28 of each cycle and rituximab IV on day 1 of event numbered cycles. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may optionally continue to receive nemtabrutinib PO QD in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy during screening and may undergo throughout the trial and PET-CT scan and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Nemtabrutinib; Procedure: Positron Emission Tomography and Computed Tomography Scan; Biological: Rituximab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Nemtabrutinib — Given PO
  Other Names: ARQ 531; ARQ-531; ARQ531; Bruton's Tyrosine Kinase Inhibitor ARQ 531; BTK Inhibitor ARQ 531; MK-1026
Procedure: Positron Emission Tomography and Computed Tomography Scan — Undergo PET-CT scan
  Other Names: PET-CT Scan; PET/CT SCAN; Positron Emission Tomography/Computed Tomography
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This phase II trial tests how well nemtabrutinib works with rituximab for the treatment of patients with mantle cell lymphoma. Nemtabrutinib is in a class of medications called kinase inhibitors. It blocks a protein called BTK, which is present on B-cell (a type of white blood cells) cancers such as mantel cell lymphoma at abnormal levels. This may help keep cancer cells from growing and spreading. Rituximab is a monoclonal antibody. It binds to a protein called CD20, which is found on B cells (a type of white blood cell) and some types of cancer cells. This may help the immune system kill cancer cells. Giving nemtabrutinib with rituximab may kill more cancer cells in patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECITVE:

I. To evaluate the efficacy (complete response rate) of nemtabrutinib and rituximab (Nem-R) in patients with treatment-naïve mantle cell lymphoma (MCL).

SECONDARY OBJECITVES:

I. To evaluate objective response rate (ORR), median progression-free survival (PFS), overall survival (OS) and duration of response (DOR).

II. To evaluate safety and tolerability of Nem-R in patients with treatment-naïve MCL.

EXPLORATORY OBJECITVES:

I. To conduct preliminary assessment of the predictive value of minimal residual disease (MRD) in MCL treated with a novel regimen.

II. To explore immune cell populations in patients treated with Nem-R. III. To explore mechanisms of resistance to Nem-R therapy in MCL. IV. To estimate the second PFS after salvage therapy for patients who progress after Nem-R therapy.

OUTLINE:

INDUCTION: Patients receive nemtabrutinib orally (PO) once per day (QD) on days 1-28 of each cycle and rituximab intravenously (IV) on days 1, 8, 15 and 22 of cycle 1 and on day 1 of subsequent cycles. Cycles repeat every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive nemtabrutinib PO QD on days 1-28 of each cycle and rituximab IV on day 1 of event numbered cycles. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may optionally continue to receive nemtabrutinib PO QD in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow biopsy during screening and may undergo throughout the trial and positron emission tomography-computed tomography (PET-CT) scan and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, then every 3 months for the first 2 years and every 6 months for the third year for patients in remission at the end of treatment or every 6 months for patients who end response follow up.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Age: ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Diagnosis of MCL established by histologic assessment including one of the following:

  * Immunohistochemistry of the biopsy
  * Flow cytometry of the biopsy
* Requiring treatment for MCL, and for which no prior systemic anticancer therapies have been received

  * Local radiotherapy not exceeding a total dose of 20 gray (Gy) at least 2 weeks prior the first dose of study therapy is allowed
* Laboratory, radiographic, physical exam findings and/or symptoms attributable to MCL.

  * Asymptomatic patients with blastoid or pleomorphic variant can be enrolled
* Radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (as defined by Lugano Classification for non hodgkin's lymphoma [NHL])
* Without bone marrow involvement: absolute neutrophil count (ANC) ≥ 1,000/mm^3, with bone marrow involvement: ANC ≥ 500/mm^3

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* Without bone marrow involvement: platelets ≥ 75,000/mm^3 with bone marrow involvement: platelets ≥ 30,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Serum creatinine ≤ 1.5 × ULN OR creatinine clearance of ≥ 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin time (PT) ≤ 1.5 × ULN, if on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, if on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Seronegative for hepatitis C virus (HCV), hepatitis B virus (HBV) (surface antigen negative) OR

  * If seropositive for HBV or HCV, nucleic acid quantitation must be performed. Viral load must be undetectable. Patients with occult or prior HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) may be included if HBV deoxyribonucleic acid (DNA) is undetectable, if they are willing to undergo DNA testing on day 1 of every cycle and every three months for at least 12 months after the last cycle of study treatment
* Participants with HIV are eligible if they meet ALL the following:

  * CD4 count > 350 cells/uL at screening
  * The HIV viral load is below the detectable level as per locally available testing
  * Are on a stable antiretroviral therapy (ART) regimen for at least 4 weeks prior to study entry

    * NOTE: ART includes drugs, which are NOT strong CYP3A4 inducers (participants receiving ART that are strong CYP3A4 inducers are not eligible to be included in the study).
  * HIV screening tests are not required unless:

    * Known history of HIV infection
    * As mandated by local health authority
  * Are compliant with their ART NOTE: If the participant has had an AIDS defining opportunistic infection in the past 12 months prior to screening, they are not eligible to be included in the study
* Person of childbearing potential (POCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Participants assigned male sex at birth:

If capable of producing sperm, the participant agrees to the following during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention. The length of time required to continue contraception for each study intervention is:

* Nemtabrutinib: 12 days
* Rituximab: 3 months
* Abstains from penile-vaginal intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agrees to remain abstinent OR
* Uses contraception as detailed below unless confirmed to be azoospermic (vasectomized or secondary to medical cause, documented from the site personnel's review of the participant's medical records, medical examination, or medical history interview) as detailed below:
* Uses a penile/external condom plus nonparticipant of childbearing potential who is not currently pregnant and should also be advised of the benefit for that partner to use an additional method of contraception, as a condom may break or leak.

  * Note: Participants capable of producing ejaculate whose partner is pregnant or breastfeeding must agree to use penile/external condom during each episode of sexual activity in which the partner is at risk of drug exposure via ejaculate.
* Contraceptive use by participants capable of producing sperm should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions are more stringent than the requirements above, the local label requirements are to be followed

  * Participants assigned female sex at birth:

A participant assigned female sex at birth is eligible to participate if not pregnant or breastfeeding, and at least one of the following conditions applies:

* Is not a person of childbearing potential (POCBP) OR
* Is a POCBP and:

  * Uses a contraceptive method that is highly effective (with a failure rate of < 1% per year), with low user dependency, or is abstinent from penile-vaginal intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention. The length of time required to continue contraception for each study intervention is:
  * Nemtabrutinib: 1 month
  * Rituximab: 12 months
  * The investigator should evaluate the potential for contraceptive method failure (ie, noncompliance, recently initiated) in relationship to the first dose of study intervention. Contraceptive use by POCBPs should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. If the contraception requirements in the local label for any of the study interventions are more stringent than the requirements above, the local label requirements are to be followed.
* Has a negative highly sensitive pregnancy test (urine or serum) as required by local regulations within 24 hours (for urine test) or 72 hours (for serum test) before the first dose of study intervention. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Abstains from breastfeeding during the study intervention period and for at least 30 days after study intervention with nemtabrutinib.
* Medical history, menstrual history, and recent sexual activity has been reviewed by the investigator to decrease the risk for inclusion of a POCBP with an early undetected pregnancy

Exclusion Criteria:

* Chronic systemic corticosteroid use > 20 mg/day of prednisone or equivalent. Patients who received corticosteroid treatment with ≤ 20 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to day 1 of cycle 1. Patients may have received a brief (≤ 14 days) course of systemic steroids (≤ 100 mg prednisone equivalent per day) prior to initiation of study therapy for control of lymphoma-related symptoms
* History of severe bleeding disorder defined as an ongoing congenital or acquired condition that leads to an increased likelihood of bleeding
* Unstable cardiac disease as defined by one of the following:

  * Acute myocardial infarction (MI) within the past 6 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Unstable angina (angina symptoms at rest) or new-onset angina (begun within the last 3 months)
* Corrected QT (QTc) prolongation (defined as a Fridericia's corrected QT interval [QTcF] > 450 msecs) or other significant electrocardiogram (ECG) abnormalities including second degree atrioventricular (AV) block type II, third degree AV block, or bradycardia (ventricular rate less than 50 beats/min)
* Positive for hepatitis C virus (HCV) virus by polymerase chain raction (PCR) at screening. Testing only required if the hepatitis (hep) C antibody is positive
* AIDS-defining opportunistic infection in the past 12 months prior to screening
* Known allergy/sensitivity (≥ grade 3) to nemtabrutinib or any of the excipients; history of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents
* Clinically significant uncontrolled illness
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection (as evaluated by the investigator) within 4 weeks prior to the first study treatment
* Primary or secondary central nervous system (CNS) lymphoma at the time of recruitment or history of CNS lymphoma
* Other active malignancy. Exceptions include malignancy treated with curative intent and no known active disease present for ≥ 2 years prior to initiation of protocol therapy; adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease; adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease; asymptomatic prostate cancer managed with "watch and wait" strategy
* POCBP: Pregnant or breastfeeding
* Patients with gastrointestinal dysfunction and/or clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea, vomiting or any other condition that will interfere significantly with drug absorption (e.g., gastric bypass surgery, gastrectomy)
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-01-08 (Estimated); Study Completion 2027-01-08 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | Up to 5.5 years
  Defined as the proportion of response-evaluable participants that achieve a best response of complete response (CR) at any time on the study prior to any disease progression or start of other anti-lymphoma therapy. Will be estimated among response-evaluable participants along with the 95% exact binomial confidence interval.

SECONDARY OUTCOMES:
Overall response rate | Up to 5.5 years
  Defined as the proportion of response-evaluable participants that achieve a best response of either CR or partial response (PR) any time on the study prior to any disease progression or start of other anti-lymphoma therapy. Will be estimated among response-evaluable participants along with the 95% exact binomial confidence interval.
Progression free survival | From start of protocol treatment to disease relapse/progression, start of other anti-lymphoma therapy, or death due to any cause, whichever occurs earlier, up to 5.5 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Overall survival | From start of protocol treatment to death due to any cause, up to 5.5 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Duration of response | From the first achievement of PR or CR to time of progressive disease, start of non-protocol anti-lymphoma therapy, or death, whichever earlier, up to 5.5 years
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation.
Incidence of adverse events | Up to 5.5 years
  Toxicities/adverse events will be recorded and severity assessment will be the National Cancer Institute Common Terminology Criteria for Adverse Events 5.0 scale. Toxicities will be summarized by time of onset, type, severity, and attribution.

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California